CLINICAL TRIAL: NCT00612209
Title: A Phase 1 Dose Escalation Study of ARQ 197 Given Twice Daily Continuously in Adult Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ARQ 197 in Adult Patients With Advanced Solid Tumors
Acronym: ARQ 197
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-103
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Cancer, Advanced Solid Tumors
Keywords: ARQ 197, advanced solid tumors, phase 1, dose escalation, pharmacodynamics, safety
MeSH Terms: conditions — Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ARQ 197

INTERVENTIONS:
Drug: ARQ 197 — Treatment with ARQ 197

SUMMARY:
This is an open label, single arm, dose escalation study of ARQ 197 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Patients will take ARQ 197 orally twice daily continuously at dose levels specified for their respective dose cohorts. The ARQ 197 starting dose will be a total daily dose of 200 mg (100 mg bid). ARQ 197 treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, dose adjustment is permitted. A treatment cycle is designed as four weeks (28 days) and will be repeated without therapy interruption.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented according to ICH GCP, the local regulatory requirements, and permission to use private health information in accordance with HIPPA prior to study-specific screening procedures
* A histologically or cytologically confirmed advanced solid tumor, including 10 patients with advanced prostate cancers in the expansion cohort.
* ≥ 18 years of age.
* Patients must have accessible tumor that is safely amenable to tumor biopsies.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors
* Tumor imageable by DCE-MRI preferably > 3cm in abdomen, pelvis, head/neck or peripheral limb (only for 12 patients undergoing MRI studies including DCE-MRI and DW-MRI in the expanded cohort)
* Karnofsky performance status (KPS) ≥ 70% or Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last ARQ 197 dose
* Females of childbearing potential must have a negative serum pregnancy test
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5.0 × ULN with metastatic liver disease
* Hemoglobin ≥ 10 g/dl
* Total bilirubin ≤ 1.5 × ULN
* Creatinine ≤ 1.5 x ULN
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L

The following inclusion criteria apply to patients with prostate cancer only:

* Histologically documented adenocarcinoma of the prostate, clinically refractory or resistant to hormone therapy, as documented by progression following castration
* PSA or radiological evidence for progressive prostate cancer
* Ongoing gonadal androgen deprivation therapy with LHRH analogues or orchiectomy. Patients who have not had an orchiectomy must be maintained on effective LHRH analogue therapy before and during the trial.
* Castrate testosterone level [< 50 ng/dL or < 2.00 nmol/L (nmol/L x 28.8 = ng/dL)]

Exclusion Criteria:

* Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks prior to first dose of ARQ 197
* Surgery within 4 weeks prior to first dose
* Known untreated brain metastases
* Pregnant or breastfeeding
* Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection)
* Unable or unwilling to swallow ARQ 197 capsules twice daily
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
* For patients undergoing magnetic resonance imaging (MRI) studies (including DCE-MRI and DW-MRI) in the expanded cohort:
* Contraindications to MRI, e.g. contraindicated metal implants
* Patients with Creatinine > x1 ULN
* Patients without antecubital fossa venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability | ARQ 197 treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met

SECONDARY OUTCOMES:
To evaluate pharmacodynamics of phosphorylated c-Met, total c-Met, apoptosis marker (TUNEL) and phosphorylated FAK in tumor tissue correlated with administration of ARQ 197. | ARQ 197 treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met
To assess the preliminary anti-tumor activity of ARQ 197. | ARQ 197 treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met
To determine the pharmacokinetic (PK) profile of ARQ 197 with continuously twice daily oral dosing schedule. | ARQ 197 treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met

CONTACTS AND LOCATIONS:
Overall Officials: Johann DeBono, MBChB, FRCP, Principal Investigator — The Royal Marsden Hospital
Locations (1):
- The Royal Marsden Hospital, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Yap TA, Olmos D, Brunetto AT, Tunariu N, Barriuso J, Riisnaes R, Pope L, Clark J, Futreal A, Germuska M, Collins D, deSouza NM, Leach MO, Savage RE, Waghorne C, Chai F, Garmey E, Schwartz B, Kaye SB, de Bono JS. Phase I trial of a selective c-MET inhibitor ARQ 197 incorporating proof of mechanism pharmacodynamic studies. J Clin Oncol. 2011 Apr 1;29(10):1271-9. doi: 10.1200/JCO.2010.31.0367. Epub 2011 Mar 7. PMID 21383285